CLINICAL TRIAL: NCT05225766
Title: Comparison of Intraoperative and Postoperative Effects of Erector Spinae Plane Block and Rectus Sheath Block
Brief Title: Comparison of Erector Spinae Plane Block and Rectus Sheath Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Emre Salman, Principal investigator, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TurkishARD
Record Dates: First submitted 2021-11-08; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Postoperative Pain, Acute
Keywords: erector spinae plane block; rectus sheath block; pain management; midline laparotomy
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESPB (Active Comparator): Erector spinae plane block
  Interventions: Other: bupivacaine
- Group RSB (Active Comparator): Rectus sheath block
  Interventions: Other: bupivacaine

INTERVENTIONS:
Other: bupivacaine — used for peripheral block

SUMMARY:
In study, The investigators aimed to compare the intraoperative and postoperative analgesic efficacy of erector spinae plane block and rectus sheath block, which investigators routinely perform in surgeries with abdominal lover midline-upper midline incision, morphine consumption with patient-controlled analgesia, as well as patient and surgeon satisfaction.

DETAILED DESCRIPTION:
Following ethics committee approval and written consent from the patients, the study was conducted on 60 patients aged between 18-75 years in American Society of Anesthesiologists (ASA) classes I-III, who were to undergo midline incisions. The demographic data of the patients were recorded and after routine monitoring and general anesthesia induction, they were divided into two groups as the ESPB group and RSB group. Hemodynamic data of all patients were recorded before induction, one minute after induction, and intraoperatively in 30-minute periods. Patient-controlled analgesia (PCA) prepared with morphine was administered to all patients. Patients' intraoperative hemodynamic data and administered opioid doses, postoperative visual analog scales (VAS) at rest and during coughing, time to first PCA dose, postoperative morphine consumption, need for rescue analgesics, duration time until first mobilization, opioid side effects, and patient and surgeon satisfaction were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years
* American Society of Anesthesiologists (ASA) classes I-III

Exclusion Criteria:

* Local anesthetic allergy
* Coagulopathy
* Injection site infection
* History of abdominal surgery
* Severe neurological or psychiatric disorder
* Severe cardiovascular disease, liver failure, renal failure (glomerular filtration rate <15 ml/min/1.73 m2)
* chronic opioid use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
intraoperative hemodynamic data and administered opioid doses | 150 minutes
  Intraoperative hemodynamic values (peripheric oxigen saturation, mean arterial pressure, heart rate) of the patients and intraoperative opioid consumption (mg) were compared.
postoperative visual analog scales at rest and during coughing | 48 hours
  Postoperatively, both coughing and resting visual analog scale values (A rating between 0 and 10 was made. 0 no pain 10 severe pain) of the patients were recorded and compared between the groups.
time to first patient controlled analgesia (PCA) dose | 48 hours
  The times when patients used the PCA device for the first time were recorded and compared between groups.
postoperative morphine consumption | 48 hours
  Total morphine (mg) consumptions used with postoperative PCA were recorded and compared between groups.
need for rescue analgesics | 48 hours
  Bolus-dose morphine administration was provided to patients with VAS ≥4 upon questioning in the clinic or in line with patients' complaints, and patients' VAS scores during the first use of PCA were recorded. It was planned for rescue analgesic to be administered in patients with VAS ≥4 despite PCA, firstly as 20 mg IV tenoxicam (Tilcotil®, Deva, Tekirdağ, Turkey), and secondly as 50 mg IV tramadol (Tramosel®, Haver, Istanbul, Turkey) if VAS was still ≥4 one hour after tenoxicam administration.
duration time until first mobilization | 48 hours
  The times until the first mobilization of the patients were recorded and it was investigated whether there was a difference between the groups in terms of mobilization times.
opioid side effects | 48 hours
  Side effects (nausea, vomiting and sedation) that may occur due to opioid use in patients were recorded. And it was investigated whether there was a difference between the groups.
patient and surgeon satisfaction | 48 hours
  Patient and surgical team satisfaction were recorded using a 5-point Likert scale (A rating of 1 to 5 was requested. 1- not at all satisfied 2- somewhat satisfied 3- undecided 4- satisfied 5- very satisfied).The difference between the groups was investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Emre SALMAN, MD, Principal Investigator — Investigator
Locations (1):
- Bursa Uludag University, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No